CLINICAL TRIAL: NCT06176157
Title: Vitamin D Supplementation in Vitamin D Deficient/Insufficient Children Oral or Parenteral! D2 or D3, A Randomized Controlled Trial.
Brief Title: Vitamin D Supplementation in Pediatrics. Oral or Parenteral! D2 or D3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Magdy Hassan Nawar, Lecturer of Pediatric Endocrinology, Faculty of Medicine, Ain Shams University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS468/2023
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D, ergochalciferol, cholecalciferol, oral, parenteral
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- oral vitamin D2 group (Active Comparator)
  Interventions: Dietary Supplement: vitamin D2, vitamin D3
- oral vitamin D3 group (Active Comparator)
  Interventions: Dietary Supplement: vitamin D2, vitamin D3
- Parenteral vitamin D2 group (Active Comparator)
  Interventions: Dietary Supplement: vitamin D2, vitamin D3
- Parenteral vitamin D3 group (Active Comparator)
  Interventions: Dietary Supplement: vitamin D2, vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D2, vitamin D3 — comparing parentral D2, D3, to oral D2, D3

SUMMARY:
A study will be performed on Vitamin D deficient/ insufficient Egyptian children to compare the efficacy of oral and parenteral forms of Ergocalciferol and cholecalciferol in raising serum 25(OH) D levels in these subjects

ELIGIBILITY:
Inclusion Criteria:

* laboratory evidence of vitamin D deficiency or insufficiency without clinical signs of rickets

Exclusion Criteria:

* vitamin D or calcium supplementation within the last 6 months before inclusion, patients with diabetes mellitus, chronic liver disease and kidney disease, congenital or rheumatic heart disease, malabsorption syndromes, thyroid disease, juvenile rheumatic diseases, or other bone disorders.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
serum 25(OH) D level after 1,2,3 months of supplementation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Nawar, Lecturer, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: Undecided
After Publishing the research individual data will be available